CLINICAL TRIAL: NCT01517061
Title: Integrative Genomic Analysis In Phantom Limb Pain
Brief Title: Genetics and Phantom Limb Pain
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120054; 12-NR-0054
Record Dates: First submitted 2012-01-24; First posted 2012-01-25 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2014-07-30

CONDITIONS: Polymorphism-Genetic; Amputation; Pain
Keywords: Phantom Limb Pain; Genetic Polymorphisms; Genetic Susceptibility; Amputation
MeSH Terms: conditions — Pain; Phantom Limb; Genetic Predisposition to Disease

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Background:

- Many people who lose a limb feel pain in the missing limb. This feeling is called phantom limb pain. Researchers do not fully understand what causes this pain. Differences in people's genes may play a role. Comparing the genes of people with and without phantom limb pain may help researchers better understand this feeling, who is likely to develop it, and how to treat it.

Objectives:

- To study whether genetic differences affect phantom limb pain.

Eligibility:

- Individuals at least 18 years of age who have lost an arm or leg at least 3 months ago.

Design:

* Participants will be screened with a medical history and physical exam.
* Participants will answer questions about how they lost the limb, and whether they feel phantom limb pain. They will also have a test to measure their sensitivity to heat and cold.
* Participants will provide a blood sample for genetic testing.

DETAILED DESCRIPTION:
Objectives:

The proposed clinical trial will investigate the role of the human genome including genetic variations and gene expression profiles on the development of phantom limb pain (PLP).

Study population:

Patients will be recruited from military personnel with major limb amputations. A total of one thousand subjects with upper or lower extremity amputations of any level will be enrolled in this study.

Design:

Eight hundred subjects with chronic PLP (PLP patient) and 200 patients without PLP (non-PLP patient) will assess the severity of their pain symptom. Each participant will undergo a routine blood draw from which DNA and RNA will be harvested.

Outcome measures:

Using Affymetrix SNP 6.0 technology, which identifies up to 1 million single nucleotide polymorphisms (SNPs) and 1 million copy number variations in the human genome, the differences in genomic variations between the PLP and the non-PLP patients will be analyzed. An extreme subset of PLP patients will be tested for their quantitative sensory function and profiled gene expression and epigenetic pattern with the Affymetrix Human Exon ST 1.0 and Illumina Genome Analyzer IIx. These integrative genomic analyses using genetic variations, gene expression and epigenetic profile could explain why some amputees experience chronic PLP and some do not. By studying these responses in patient samples, we will evaluate the role of genomic factors in PLP. SNP frequencies, gene expression and epigenetic profiles between PLP and non-PLP groups will be analyzed.

ELIGIBILITY:
* INCLUSION CRITERIA:

PLP GROUP:

* at least 18 years of age
* Single or multiple upper and/or lower limb amputation
* At least three months post-amputation
* Ability to follow study instructions in English
* Currently present on-going PLP for at least one month and at least 3 times per week

NON PLP GROUP:

-same with PLP group except:

--Experienced PLP less than 10 times total and/or for less than two weeks

EXCLUSION CRITERIA:

BOTH PLP AND NON-PLP GROUPS:

* Chronic systemic disease which might affect pain sensitivity and ability to participate in this study s blood draw
* Any disease (such as hemophilia) or medication regimen (such as warfarin) increasing hemorrhage that would make a blood draw dangerous or inadvisable for the subject
* Known uncontrolled systemic diseases; known cancer not in remission, known on-going infection, lupus, kidney disease requiring dialysis, any other systemic disease which might affect ability to participate in this study s blood draw
* Inability to provide his/her own informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01-03; Study Completion 2014-07-30

PRIMARY OUTCOMES:
SNP frequency between PLP and non-PLP group

SECONDARY OUTCOMES:
Gene expression profile between PLP and non-PLP group
Epigenetic profile between PLP and non-PLP group

CONTACTS AND LOCATIONS:
Overall Officials: Hyungsuk Kim, D.D.S., Principal Investigator — National Institute of Nursing Research (NINR)

REFERENCES:
- [Background] Weinstein SM. Phantom limb pain and related disorders. Neurol Clin. 1998 Nov;16(4):919-36. doi: 10.1016/s0733-8619(05)70105-5. PMID 9767070
- [Background] Sherman RA, Sherman CJ. Prevalence and characteristics of chronic phantom limb pain among American veterans. Results of a trial survey. Am J Phys Med. 1983 Oct;62(5):227-38. PMID 6624883
- [Background] Montoya P, Larbig W, Grulke N, Flor H, Taub E, Birbaumer N. The relationship of phantom limb pain to other phantom limb phenomena in upper extremity amputees. Pain. 1997 Aug;72(1-2):87-93. doi: 10.1016/s0304-3959(97)00004-3. PMID 9272791